CLINICAL TRIAL: NCT02984046
Title: Acute Bronchiolitis and Severity Markers: Interest in Protein CC16
Acronym: CC16
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0294; 2015-A01587-42 (Other: 2015-A01587-42)
Record Dates: First submitted 2016-11-28; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Bronchiolitis
Keywords: Acute bronchiolitis; RSV; CC16; SP-D; sRAGE; Severity; Biomarkers

ARMS (1):
- acute bronchiolitis (Experimental): Prospective, monocentric, case-control and study Primary end-point: correlation between serum CC16 level and severity of the bronchiolitis, evaluated by a clinical scoring system
  Interventions: Drug: Protein CC16

INTERVENTIONS:
Drug: Protein CC16

SUMMARY:
Acute bronchiolitis is a common viral infection in infants mainly due to RSV and rhinovirus.

Biomarkers can be useful for predicting its severity. The serum CC16 is a marker of epithelial aggression. Its rate increase during RSV bronchiolitis in infants less than 7 months. It could be an early predictive biomarker of the severity of acute bronchiolitis, and secondarily for the development of asthma.

Two other markers of airway aggression seem to increase during acute bronchiolitis: serum SP-D protein and serum soluble receptor sRAGE.

DETAILED DESCRIPTION:
Prospective, monocentric, case-control and study Primary end-point: correlation between serum CC16 level and severity of the bronchiolitis, evaluated by a clinical scoring system established at the time of the admission in Paediatric Emergency Unit. Secondary end-points: correlation with urinary CC16; correlation with risk factors for bronchial epithelial aggression, viruses, immediate morbidity and mortality. Study of serum SP-D and sRAGE levels.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 1 year old hospitalized for acute bronchiolitis

Exclusion Criteria:

* Broncho dysplasia
* Preterm under 34 weeks
* Cystic fibrosis
* Immune deficiency
* Suspicion of primary ciliary dyskinesia
* Congenital heart disease
* Acute renal failure

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-08 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Serum CC16 rate | at day 1

SECONDARY OUTCOMES:
Urinary CC16 rate | at day 1
SP-D rates | at day 1
sRAGE rates | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: André LABBE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France